CLINICAL TRIAL: NCT03912922
Title: SIT LESS 4: How Does Reducing Sitting Time Improve Glucose and Lipid Metabolism? A Study to Identify Underlying Mechanisms
Brief Title: SIT LESS 4: How Does Reducing Sitting Time Improve Glucose and Lipid Metabolism?
Acronym: SITLESS4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Dutch Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: NL62413.068.17
Record Dates: First submitted 2019-04-03; First posted 2019-04-11 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Overweight and Obesity
Keywords: insulin sensitivity; sitting time
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sit regime (Experimental): Subjects will follow the sit regime during four days. Each day consists of 14 hours sitting, 1 hour walking and 1 hour standing and 8 hours sleeping.
  Interventions: Other: Activity regime
- Sit less regime (Experimental): Subjects will follow the sit less regime during four days. Each day will consist of 9 hours sitting, 3 hours walking, 4 hours standing and 8 hours sleeping.
  Interventions: Other: Activity regime
- Exercise regime (Experimental): Subjects will follow the exercise regime during four days. Each day will consist of 13 hours sitting, 1 hour walking, 1 hour standing, 1 hour exercise and 8 hours sleeping. The cycle session will be at approximately 60% maximal power. Exact cycling intensity and duration will be calculated to ensure equal total energy expenditure between the sitting less and the exercise regime.
  Interventions: Other: Activity regime

INTERVENTIONS:
Other: Activity regime — Activity regime of 4 days followed by a test day.

SUMMARY:
Research has shown that replacing sitting time with low intensity physical activity (such as slowly walking and standing) has beneficial effects on metabolic health, like insulin sensitivity, comparable to improvements after sitting all day in combination with 1h streneous exercise.

The main objective of this study is to investigate the underlying mechanisms responsible for improved insulin sensitivity after 4 days of sitting less compared to sitting and exercise in healthy obese women. Our secondary objective is to investigate the effects of sitting less on cardio metabolic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Caucasian
* Postmenopausal women
* Aged 45-70 years at start of the study
* Body mass index (BMI) 25 - 35 kg/m2
* Stable dietary habits (no weight loss or gain >5kg in the past 3 months)
* Sedentary lifestyle (not more than 2,5 hours of exercise per week in the past 3 months)

Exclusion Criteria:

* Not able to complete the sitless try-out day according to the protocol
* Active diseases (cardiovascular, diabetes, liver, kidney, cancer or other)
* No use of medication interfering with investigated study parameters (as determined by responsible physician)
* Alcohol consumption of >2 servings per day
* Smoking in the past 6 months
* Participation in another biomedical trial which may have an effect on insulin sensitivity less than one month before the start of the study (screening visit)
* Mental or physical disability which interferes with physical activity
* Subjects with contra-indications for magnetic resonance imaging (MRI)
* Reported participation in night shift work 2 weeks prior to the start of the study (screening visit) and during study participation. Night work is defined as working between midnight and 6.00 AM.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Day 5 of intervention period
  2-step hyperinsulinemic euglycemic clamp

SECONDARY OUTCOMES:
ex vivo skeletal muscle mitochondrial respiration | Day 5 of intervention period
  oxygraph
substrate oxidation | Day 5 of intervention period
  indirect calorimetry RER
Intrahepatic lipid content | Day 5 of intervention period
  magnetic resonance spectroscopy
Blood pressure | Day 5 of intervention period
  average resting blood pressure over 30 minutes
Plasma cardio metabolic markers | Day 5 of intervention period
  endothelial dysfunction score (average Z-score of log transformed plasma sVCAM1, sICAM1 and sE-selectin)

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Derived] Remie CME, Janssens GE, Bilet L, van Weeghel M, Duvivier BMFM, de Wit VHW, Connell NJ, Jorgensen JA, Schomakers BV, Schrauwen-Hinderling VB, Hoeks J, Hesselink MKC, Phielix E, Houtkooper RH, Schrauwen P. Sitting less elicits metabolic responses similar to exercise and enhances insulin sensitivity in postmenopausal women. Diabetologia. 2021 Dec;64(12):2817-2828. doi: 10.1007/s00125-021-05558-5. Epub 2021 Sep 12. PMID 34510226